CLINICAL TRIAL: NCT01470638
Title: Analyzes of Cerebrospinal Fluid in Autoimmune Systemic Diseases
Brief Title: A Study of Flt3-Ligand Levels in Sjögrens Syndrome
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Flt3-L SS
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Sjogrens Syndrome
Keywords: Flt3-L; CSF
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, cerebrospinal fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to correlate levels of Flt3-ligand in Cerebrospinal Fluid (CSF) and serum to markers for inflammation and degeneration in patients with primary Sjogrens syndrome.

DETAILED DESCRIPTION:
The study aims to correlate levels of Flt3-ligand in CSF and serum to markers for inflammation and degeneration in patients with primary Sjogrens syndrome.

ELIGIBILITY:
Inclusion Criteria:

* fulfill the ACR-criteria for primary Sjogrens syndrome,
* age above 18 years old

Exclusion Criteria:

* other CNS-disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The rheumatology clinic at Sahlgrenska University hospital, Gothenburg, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Correlate levels of Flt3-ligand in Cerebrospinal Fluid (CSF) and serum to markers for inflammation and degeneration in patients with primary Sjogrens syndrome | June 2009 - June 2015

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Rheumatology, Sahlgrenska University Hospital, Gothenburg, Sweden